CLINICAL TRIAL: NCT03846375
Title: Emotional Dysregulation in Para-suicidal Behavior: Effects of Dialectical Behavioral Therapy on Emotional Processing, a Triangulation Approach
Brief Title: Emotional Dysregulation in Para-suicidal Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1554/REK-C
Record Dates: First submitted 2018-11-27; First posted 2019-02-19 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-11

CONDITIONS: Self Harm; Suicide, Attempted; Emotional Instability; Borderline Personality Disorder
Keywords: Emotional Dysregulation; Emotional regulation; Dialectical Behavioral Therapy; para-suicidal behavior
MeSH Terms: conditions — Self-Injurious Behavior; Suicide, Attempted; Borderline Personality Disorder; Emotional Regulation | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: Naturalistic cohort pre-post study. However, we also include a matched control sample of healthy controls to complete the battery of measurements at pre-intervention assessments.
Masking Description: Control group only at pre-intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants in DBT (Experimental): Psychotherapy: The participants will be given standard DBT treatment.
  Interventions: Behavioral: Psychotherapy; Other: Pre-intervention testing
- Control Group (Other): Control Group at preintervention.
  Interventions: Other: Pre-intervention testing

INTERVENTIONS:
Behavioral: Psychotherapy — DBT is a well-established treatment for recurrent self-harm and suicidal thoughts. The program is principle-based, but the skills training follow a manualized curriculum.
  Arms: Participants in DBT
Other: Pre-intervention testing — Pre-intervention testing for baseline measures.

SUMMARY:
This is a naturalistic cohort pre-post study investigating aspects of emotional processing and how possible changes in emotional processing is related to the successful treatment of non-suicidal self-injury and suicidal ideation in a program of Dialectical Behavior Therapy. In addition we wish to identify to what extent the intensity and frequency of non-suicidal self-injury and suicidal ideation is related to difficulty in emotion regulation, as indicated by self-report measures and psychophysiological measures.

DETAILED DESCRIPTION:
This naturalistic pre-port study tests if Dialectical Behavior Therapy (DBT) - an established therapy addressing emotion regulation and reduction of non-suicidal self-injury and suicidal ideation - result in increased emotion regulation capacity, indicated by lowered heart rate variability (HRV) and self-report measures. The study will also test the impact of DBT on lowered non-suicidal self-injury and suicidal ideation. Standard Clinical symptom scales will be included in order to control for anxiety, depression, as well as a measure of impulsivity, which is common co-morbidities.

Since DBT was developed in the 80ies, DBT has gathered increased empirical support as a treatment that reduce suicidality, para-suicidal behavior, experienced and expressed anger, and increased social skills. In DBT, emotional dysregulation is assumed to arise from a combination of biological vulnerability and living in an invalidating environment.

Self-harm and chronic suicidality is considered to be an emotion regulation strategy. In DBT, the ability to regulate emotions adaptively requires a set of skills; the ability to experience emotions, the ability to label emotions, and the ability to modulate stimuli that serve to reactivate negative or positive emotions. In the absence of these skills, or instances where the individual is hindered from applying them, more maladaptive behavior is learned and applied. Individuals that engage in non-suicidal self-injury often report greater emotion dysregulation than those without an non-suicidal self-injury history. Such behavior can e.g. be self-inflicted harm, cutting, burning, or hitting , and/or suicidal ideation. Non-suicidal self-injury is viewed as a learned emotion regulation strategy; because such behavior instantly can decrease the experience of negative affect. Therapies that focus on increasing adaptive emotion regulations skills have demonstrated reduced non-suicidal self-injury and suicidal ideation.

The physiological manifestations of emotions rely on an activation of the Autonomic Nervous System. The individual experience of emotions is reciprocally related to the continuously changing levels of physiological arousal. The functioning of this system is in turn related to adapting to environmental demands. A well established measure of Autonomic Nervous activity is variation in inter-beat-intervals due to respiratory influence on heart rate, i.e. respiratory sinus arrhythmia, which is predominately a parasympathetic related innervation of the heart. Hence, HRV is considered a psychophysiological index of emotion regulation abilities. HRV is considered an index of the nervous system's ability to flexibly adapt to changing environmental demands and is considered a biological index of emotion regulation.

We include a matched control sample of healthy controls to complete the battery of measurements at baseline assessment of emotion regulation functions (pre-intervention assessments). This will give the opportunity to characterize the group of patients with non-suicidal self-injury and suicidal ideation included in the current planned study in relation to previous research findings of the same functions in samples of patients with non-suicidal self-injury and suicidal ideation. The combination of clinical, cognitive and psychophysiological measures is a unique feature of this study, and will provide new information regarding the mechanisms underpinning clinical change following DBT, and possibly validate heart rate variability as a possible psychophysiological outcome measure for studies on treatment for non-suicidal self-injury and suicidal ideation.

Statistical analyses Multilevel between-group analyses will be conducted to test for the between-group effects on the measures at baseline. Furthermore, a multiple regression analyses, so that dimensional variables can be included as independent variables in the model, for the pre and post measures. Regression analyses also allow for adjusting for the effects of possible confounders on the outcome measures, such as age, sex, and intensity of depressive symptoms. Furthermore, bootstrapping analysis will be conducted to examine moderator and mediator effects on the outcome measures. Interpretation of the strength of experimental effects will be guided by the use of effect size statistics. Baseline measures of demographics, life experiences, and symptoms may also be used to predict outcomes or as covariates in our analyses.

ELIGIBILITY:
Inclusion Criteria Patients:

* Patients with non-suicidal self-injury and/or suicidal ideation that undergo standard clinical outpatient DBT treatment will be recruited.

Exclusion Criteria Patients:

* Lack of informed consent

Exclusion Criteria Healthy Controls:

* Lack of informed consent
* former or current neurological conditions
* severe psychiatric illness
* cardiac conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Change in intensity of Suicidal thoughts. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  Intensity of suicidal thoughts on a likert scale from 0 - 5 the last week.
Change in frequency of suicidal thoughts. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  Frequency of suicidal thoughts, that is the number of suicidal thoughts the last week.
Change in frequency of non-suicidal self-injury. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  The frequency of non-suicidal self-injury the last week.
Change in the intensity of impulse to non-suicidal self-injury. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  The intensity in the impulse to non-suicidal self-injury on a likert scale from 0 - 5, the last week.
Change in Heart rate variability . | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  Heart rate variability is considered an index of the nervous system's ability to flexibly adapt to changing environmental demands and is considered a biological index of emotion regulation.
Change in self reported emotion regulation ability through Difficulties in Emotion Regulation Scale. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  It is a 36 item questionnaire designed for measuring six facets of difficulties in emotion regulation. The response is give in the from of a rating of 5 point likert scale from 1 ("almost never" to 5 ("almost always). Total score range: 36- 180. It includes the following sub-scales: 1. Nonacceptance of emotional responses, 2. Difficulties engaging in goal directed behavior, 3. Impulse control difficulties, 4. Lack of emotional awareness, 5. Limited access to emotion regulation strategies, 6. Lack of emotional clarity.

SECONDARY OUTCOMES:
Change in self reported ability to be mindful through the Five Facet Mindfulness Questionnaire. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  The Five Facet Mindfulness Questionnaire is a 39-item self-report questionnaire that assesses various components of mindfulness. Each item is rated on a 1 to 5 scale with 1=never or very rarely true and 5=very often or always true; responses are summed and then divided by 39 (the number of items). The higher score represents a more mindful attitude in daily life.The total score is a aggregate of the following sub-scales: (1) "observe" (the ability to ve aware of the surroundings and inner experiences, (2) describe (the ability to describe inner experiences, (3) act aware ( being aware and present, (4) non-judge (ability to experience with acceptance, and (5) non-react (being non-reactive excessively to inner experience).
Change in self reported self-compassion through the Self-compassion Scale. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  The Self-compassion Scale questionnaire consists of 26 items. Items are rated on a five-point Likert-type scale from 1 ("almost never") to 5 ("almost always").
  Highest possible score is 130. High score indicate ability to be self-compassionate.
Change in ability to experience and verbalise emotions through Toronto Alexithymia Scale 20. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  The Toronto Alexithymia Scale 20 is a 20-item self-report questionnaire consisting of three sub-scales; 1) Difficulty Identifying feelings, 2) Difficulty Describing Feelings, and 3) Externally-oriented Thinking. The full scale range is 20-100, higher scores indicate higher problems in experiencing and verbalizing emotions, i.g. alexithymia. Subscales are summed to compute a total score Scores between 52 and 60 indicate moderate alexithymia; scores 61 and higher indicate high alexithymia.
Change in anxiety symptoms through the Beck Anxiety Inventory. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  The Beck Anxiety Inventory is a 21-item self-report inventory that measures level of anxiety during the past week. Answer being scored on a scale value of 0 (not at all) to 3 (severely). Above 30 indicate severe anxiety, below 21 indication of low og no anxiety.
Change in depressive symptoms through the Beck Depression Inventory. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  Beck Depression Inventory is a 21-item self-report inventory that measures level of depression and is a widely applied measure of depression. Highest possible score is 64. Above 25 indicates severe depressive symptoms, below 9 no depressive symptoms.
Change in impulsivity through The Barratt Impulsiveness Scale. | Time points will be baseline, week 16, week 32 and at completion of the DBT program, an average of 1 year.
  The Barratt Impulsiveness Scale is a questionnaire designed to assess the personality / behavioral construct of impulsiveness is composed of 30 items describing common impulsive or non-impulsive (for reversed scored items) behaviors and preferences .

OTHER OUTCOMES:
International Neuropsychiatric Interview. | Time points will be baseline and at completion of the DBT program, an average of 1 year.
  The International Neuropsychiatric Interview is a semi-structured diagnostic interview is a structured interview to evaluate the presence of current psychiatric disorders in children, based on 10th revision of the International Statistical Classification of Diseases and Related Health Problems and Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V). The results will be combined to one binary total score 0 (no disorder) and 1 (current disorder).
Change in the presence of personality disorders through the Structured Clinical Interview for DSM-IV Axis II. | Time points will be baseline and at completion of the DBT program, an average of 1 year.
  A semi-structured diagnostic interview used to assess personality disorders according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV). The interview covers all ten DSM-IV personality disorders (antisocial, avoidant, borderline, dependent, histrionic, narcissistic, obsessive-compulsive, paranoid, schizoid and schizotypal), personality disorder not otherwise specified, and is used to make personality disorder diagnoses either dimensionally or categorically (present-absent). The instrument will applied dimensionally with scores ranging from 0 to 9. Higher score indicate the presence of personality traits.
Change in every day functioning through the Global Assessment of Functioning. | Time points will be baseline and at completion of the DBT program, an average of 1 year.
  Global Assessment of Functioning is a numeric scale used to rate subjectively the social, occupational, and psychological functioning of an individual his or her day-to-day life on a scale of 0 to 100. High score indicate high functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Berge Osnes, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bjørgvin DPS, Bergen, Norway